CLINICAL TRIAL: NCT06849895
Title: Real-World Study of Myopia Prevention and Control in Children: a Prospective Cohort Study
Brief Title: Real-World Study of Myopia Prevention and Control in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Other Study IDs: SIGCMIPCA-2024
Record Dates: First submitted 2025-02-13; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Myopia; Refractive Errors; Children; Cohort
Keywords: myopia; premyopia; outdoor activities; myopia prevention; myopia control; children; compliance; defocus optical lenses
MeSH Terms: conditions — Myopia; Refractive Errors; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Sufficient hyperopia reserve: Cycloplegic spherical equivalence is higher than the recommended values and falls within the normal range for the corresponding age group.
- Relative insufficiency in hyperopia reserve: Cycloplegic spherical equivalence is greater than +0.75 diopters but below the recommended value for the corresponding age group.
- Premyopia: -0.50 diopters < cycloplegic spherical equivalence ≤ +0.75 diopters
- Myopia: Cycloplegic spherical equivalence ≤ -0.50 diopters

SUMMARY:
This prospective, school-based cohort study aims to enroll approximately 15,000 primary school students from multiple districts in Shanghai, China and to observe the outcomes on myopia prevention and control in children with varying refractive status (including sufficient hyperopia reserve, relative insufficiency in hyperopia reserve, pre-myopia and myopia) who are exposed to a school-based categorized and integrated interventions strategy in real-world settings.

The primary objective of this study is to observe the change in the incidence and prevalence of myopia as well as the the progression of myopia among primary school students population under a school-based interventions, including increasing outdoor activities and wearing special designed optical lenses. The second objective is to identify factors influencing the outcomes and assess the compliance of different intervention methods. Additionally, a cost-effectiveness analysis will be conducted to assess the implementation process, providing technical solutions and operational models for wider application.

ELIGIBILITY:
Inclusion Criteria:

1. All students from the enrolled schools;
2. Participants must be able to cooperate with and complete all required ophthalmic examinations;
3. Written informed consent must be obtained from their parents or legal guardians.

Exclusion Criteria:

1. Ocular abnormalities (e.g., strabismus, amblyopia, or other significant eye diseases);
2. Systemic diseases that may affect ocular health;
3. Current participation in other myopia intervention programs.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All students in the enrolled schools can participate in the project and receive tiered interventions after obtaining informed consent from their guardians. After professional examination, students with conditions such as strabismus, amblyopia, other significant ocular abnormalities, systemic diseases, or those currently undergoing other myopia interventions will generally not be fitted with specially designed myopia control spectacles.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Myopia incidence | Assessed at 12 months, 24 months, and 36 months post-baseline.
  Myopia incidence
Myopia progression | Assessed at 12 months, 24 months, and 36 months post-baseline.
  Myopia progression in myopic participants

SECONDARY OUTCOMES:
Myopic shift | Assessed at 12 months, 24 months, and 36 months post-baseline.
  Change of spherical equivalence and axial length

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided